CLINICAL TRIAL: NCT04365699
Title: A Single-center Registry and Embedded Interventional Study of the Effects of COVID-19 With and Without Treatment With AT-001 on Cardiac Structure and Function in Patients Hospitalized for Management of COVID-19 Infection
Brief Title: Cardiovascular Effects of COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-00416
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — caficrestat

STUDY DESIGN:
Intervention Model Description: All subjects hospitalized with COVID-19 infection hospitalized will be enrolled in the registry; a subgroup meeting specific entry criteria listed below will be enrolled in the open-label interventional trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Interventional Patients: AT-001 (Experimental): AT-001 1500 mg (3 capsules) were administered by mouth twice daily for up to 14 days
  Interventions: Drug: AT-001
- Control Match Group 1 (No Intervention): Matched control from a contemporaneous de-identified registry of hospitalized patients with clinical COVID-19 diagnosis at the same institution was selected. The first matching approach selected all subjects with diabetes mellitus and hypertension, and available data to match participants who received AT-001 for gender, age group (in bins of 5 years), weight, and C-reactive protein (CRP) value at the time of hospital admission.
- Control Match Group 2 (No Intervention): Matched control from a contemporaneous de-identified registry of hospitalized patients with clinical COVID-19 diagnosis at the same institution was selected. The second matching approach selected all subjects in the registry with diabetes mellitus and available data to match participants who received AT-001 for gender, age group (in bings of 5 years), and weight (+/- 0.5 kgs).

INTERVENTIONS:
Drug: AT-001 — Investigational novel Aldose Reductase Inhibitor (ARI) Product: AT-001 500mg capsule for oral administration Dosage: 1,500mg (3X500mg capsules) twice daily Mode of Administration: Oral Up to 14 days per discretion of the investigators and treatment team
  Arms: Interventional Patients: AT-001

SUMMARY:
Cardiometabolic disease may confer increased risk of adverse outcomes in COVID-19 patients by activation of the aldose reductase pathway, a trigger of the inflammatory cascade. The study team hypothesizes that aldose reductase inhibition with AT-001 (caficrestat) might represent a novel therapeutic approach to reduce inflammation and risk of adverse outcomes in diabetic patients with COVID-19.

An open-label pilot study to assess safety, tolerability and efficacy of AT-001 in hospitalized COVID-19 patients with history of diabetes mellitus and heart disease will be conducted. Eligible participants will be treated with AT-001 1500 mg twice daily for up to 14 days. Safety, tolerability, survival and length of hospital stay data were compared with matched controls from a contemporaneous registry of COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria

Registry Study: In order to be eligible to participate in the registry study, an individual must meet all of the following criteria:

1. Age ≥18 years of age
2. Hospitalized at one of the participating NYULH locations
3. Confirmed COVID-19 infection

Interventional Study: In order to be eligible to participate in the registry study, and individual must meet all of the inclusion criteria of the registry study plus the following criteria:

1. Hospitalized at NYU Tisch
2. History of diabetes mellitus or blood glucose measurement >126 mg/dl AND EITHER
3. History of hypertension and/or ischemic heart disease and/or heart failure OR
4. Other co-morbid condition that in the opinion of the PI increases risk of heart or lung injury related to the aldose reductase pathway

Exclusion Criteria

Registry Study: An individual who meets any of the following criteria will be excluded from participation in the registry study:

1. Persons who have opted out of research participation at NYU
2. Pregnancy

Interventional study: An individual who meets any of the following criteria will be excluded from participation in the interventional study:

1. Persons who have opted out of research participation at NYU
2. Pregnancy
3. Women of childbearing potential
4. Breast-feeding women
5. Participation in another investigational drug protocol within previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Katz, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to Stuart.Katz@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Requests may be directed to Stuart.Katz@nyulangone.org.

RESULTS

PARTICIPANT FLOW:
Groups:
- Interventional Patients: AT-001: Patients enrolled in registry from NYU Langone Tisch Hospital with history of diabetes mellitus and/or acute hyperglycemia (any glucose measurement >200 mg/dl) and evidence of acute or chronic heart disease. This subset will receive Standard of Care + AT-001.
  AT-001: Investigational novel Aldose Reductase Inhibitor (ARI) Product: AT-001 500mg capsule for oral administration Dosage: 1,500mg (3X500mg capsules) twice daily Mode of Administration: Oral Up to 14 days per discretion of the investigators and treatment team
Period: Overall Study
Arm/Group | Interventional Patients: AT-001 | Control Match Group 1 | Control Match Group 2
Started | 10 | 16 | 55
Completed | 8 | 11 | 40
Not Completed | 2 | 5 | 15
Not completed — Death | 2 | 5 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interventional Patients: AT-001 | Control Match Group 1 | Control Match Group 2 | Total
Number analyzed (Participants) | 10 | 16 | 55 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (6.6) | 65 (7.7) | 64.5 (5.3) | 64.8 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 11 | 15
  Male | 8 | 14 | 44 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 16 | 55 | 81
Region of Enrollment [Number; unit: participants]
  United States | 10 | 16 | 55 | 81

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay (LOS)
Description: Data collection from medical chart review
Time Frame: Day 45
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Interventional Patients: AT-001 | Control Match Group 1 | Control Match Group 2
Number analyzed (Participants) | 10 | 16 | 55
days | 5 [4 to 29] | 10 [5 to 20] | 25 [16 to 36]

2. Primary Outcome: Percentage of Participants Who Died
Description: Data collection from medical chart review
Time Frame: Day 45
Measure: Number; unit: percentage of participants
Arm/Group | Interventional Patients: AT-001 | Control Match Group 1 | Control Match Group 2
Number analyzed (Participants) | 10 | 16 | 55
percentage of participants | 20 | 31.3 | 27.3

ADVERSE EVENTS:
Time Frame: 45 days
Arm/Group | Interventional Patients: AT-001 | Control Match Group 1 | Control Match Group 2
All-Cause Mortality (participants affected / at risk) | 2/10 | 5/16 | 15/55
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/16 | 0/55
Other Adverse Events (participants affected / at risk) | 3/10 | 0/16 | 0/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interventional Patients: AT-001 (N=10) | Control Match Group 1 (N=16) | Control Match Group 2 (N=55)
Nausea / Upset GI (Gastrointestinal disorders) | 2 | 0 | 0
Localized Skin Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT04365699/Prot_SAP_001.pdf